CLINICAL TRIAL: NCT00102115
Title: Phase 1 Dose Ranging Study to Evaluate Safety and Tolerability of Talaporfin Sodium (LS11) Photodynamic Therapy in Subjects With Advanced Age-Related Macular Disease
Brief Title: Study of Talaporfin Sodium Photodynamic Therapy to Treat Advanced Age Related Macular Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Light Sciences LLC (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LSCOR-001
Record Dates: First submitted 2005-01-21; First posted 2005-01-24 (Estimated); Last update posted 2010-03-12 (Estimated); Status verified 2005-12

CONDITIONS: Macular Degeneration; Choroidal Neovascularization
Keywords: Macular disease; Wet AMD; AMD; Age-Related Macular Disease; PDT; Photodynamic Therapy
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — Talaporfin; Photochemotherapy

INTERVENTIONS:
Drug: Talaporfin Sodium (LS11) Photodynamic Therapy (PDT)

SUMMARY:
The purpose of this study is to determine the safety and tolerability of Talaporfin Sodium (LS11) Photodynamic Therapy in patients with late stage Age-Related Macular Disease (AMD).

DETAILED DESCRIPTION:
This Phase 1 study is a safety and tolerability investigation of LS11 photodynamic therapy in subjects with persistent leaking neovascular membranes in patients with AMD who have a visual acuity of 20/200 or less. This is a sequential group dose escalation trial with the cohorts defined by increasing the light dose. Within each light-dose cohort, three (3) subjects will be treated at a drug dose of 0.2 mg/kg or 0.5 mg/kg.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 or older
* Subject is able to sign informed consent
* Ability to complete 6 month trial
* Present with advanced AMD and persistently leaking CNV
* Adequate hematologic, renal and liver function
* Negative pregnancy test
* Subject is able to safely undertake all protocol directed instructions
* Visual acuity of 20/200 (logMAR 1.0)(6/60) or worse

Exclusion Criteria:

* Concomitant eye disease in eye to be treated
* Prior ocular radionuclide treatments
* Known allergic or hypersensitivity reactions to light and/or fluorescein and iodine or shellfish
* History of investigational drug or therapy including biologics within 30 days prior to the study drug dosing
* Women who are pregnant or lactating, or women of childbearing years not taking adequate contraception precautions
* History of porphyria, systemic lupus erythematosus, or xeroderma pigmentosum
* History of clinically significant cardiovascular abnormalities, including myocardial infarction in the past 6 months, uncontrolled arrhythmias, uncontrolled congestive heart failure
* Concomitant use of other drugs known to produce skin photosensitivity, e.g. tetracycline, sulfonamides, phenothiazines, sulfonylureas, thiazide diuretics and griseofulvin, St. John's Wort
* Subjects with high or pathological myopia with an axial length > 26mm or a refractive error of >/= -8.00D
* Subjects with glaucoma and vision loss in either eye
* Subject with a history of other choroidal leakage, e.g. histoplasmosis
* Subjects with significant media opacity
* Subjects diagnosed with diabetic retinopathy
* Subjects who have had eye surgery within the past 3 months
* Subjects who have received PDT treatment for AMD in the treatment eye
* Any disease or condition that the sponsor or the investigator believes will impact the subject's ability to adhere to the study schedule
* Subjects participating in any concurrent trial

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27
Dates: Start 2004-12; Study Completion 2006-01

PRIMARY OUTCOMES:
Cessation of leakage from choroidal neovascularization (CNV) of subjects with late stage AMD

SECONDARY OUTCOMES:
Changes in visual performance

CONTACTS AND LOCATIONS:
Overall Officials: Gary Krasner, PhD, Study Director — Light Sciences LLC
Locations (1):
- Texas Retina, Dallas, Texas, United States